CLINICAL TRIAL: NCT03965286
Title: Effect of Direct AntiViral Drugs of Chronic HCV on eGFR in Assuit Universiry Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moamen mohey AbdElhamid, Resident doctor, Assiut University
Other Study IDs: DAAs on eGFR
Record Dates: First submitted 2019-05-19; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Antiviral Drug
MeSH Terms: interventions — ledipasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic HCV will be on direct antiviral drugs: is defined as the presence of detectable viral replication for at least six months diagnosed by quantitative HCV RNA polymerase chain reaction (PCR)
  Interventions: Drug: DAAs

INTERVENTIONS:
Drug: DAAs — Daily fixed-dose combination of ledipasvir (90 mg)/sofosbuvir (400 mg) 12 weeks Daily simeprevir (150 mg) plus sofosbuvir (400 mg) 12 weeks Daily daclatasvir (60 mg) plus sofosbuvir (400 mg) 12 weeks Daily fixed-dose combination of paritaprevir (150 mg)/ritonavir (100 mg)/ombitasvir (25 mg) with dasabuvir (600 mg) 12weeks
  Other Names: ledipasvir/sofosbuvir/daclatasvir

SUMMARY:
1. evaluation of glomerular filtration rate(eGFR)changes during HCV treatment with direct antiviral drugs according to 2018 guideline.
2. TO estimate the frequency of renal impairment by direct antiviral drugs By detection of any changes in e GFR.
3. Assessment The Renal safety during HCV treatment with direct antiviral drugs according to 2018 guideline.
4. To clarify the importance of laboratory and other modalities in detection and estimation of frequency of renal impairment by direct antiviral drugs according to 2018 guideline.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) has an estimated global prevalence of 2%-3% with 130-170 million people infected with HCV.(1) HCVcauses chronic inflammation of the liver leading to chronic hepatitis, which can advance to liver cirrhosis and hepatocellular carcinoma and significant extrahepatic complications.(2) Additionally, HCV has been shown to have a significant negative effect on apatient's overall quality of life, including decreased work hours and productivity and increased healthcare costs.(3) Cirrhosis and hepatocellular carcinoma related to HCV infection represent the most common indications for liver transplantation duo to poor treatment options.(4) Until recently, interferon-based treatments were thebackbone of HCV treatment options.(5) Unfortunately,therapy was only modestly effective and associatedwith significant side effects.(6) Therefore, research has focused on HCV eradication using oral antiviral therapy.

Recent clinical studies have demonstrated efficacy using the nucleotide analogue inhibitor sofosbuvir(Sovaldi; Gilead Sciences, Inc., Foster City, CA) as the backbone in treatment of non transplant and post transplant recurrent HCV.(7) Both the ION-1 and ION-2 trials demonstrated nearly 99% efficacy in the treatment ofnontransplant, noncirrhotic HCV patientsusing sofosbuvir in a fixed-dose combination with theNS5A inhibitor ledipasvir (Harvoni, Gilead Sciences,Inc.), both with and without ribavirin.(8,9) The side effect profile of ledipasvir/sofosbuvir (LDV/SOF) hasbeen relatively mild and the drug has been well tolerated in trials, especially compared with previous interferon-based regimens.

The ION trials report that LDV/SOF therapy was primarily complicated by headaches or fatigue inapproximately 10% of patients. Less frequently, patients experienced rashes, nausea, diarrhea, and insomnia.Serious side effects, such as nephrotoxicity, were not demonstrated by the ION-1 and ION-2 trials; however, these trials were conducted in a controlled clinical setting with rigorous exclusion criteria. Such trials are not always entirely reflective of the general patient population. Early data suggest possible risk of renal impairment during treatment with the use of direct antiviral drugs(10) this study is about renal safety and changes in eGFR in patients with chronic HCV undergoing direct acting antiviral therapy according to 2018 guideline.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C virus patients will be on direct antiviral therapy .

Exclusion Criteria:

* patients with DM ,HTN ,CKD,Autoimmune Diseases Patients with kidney injury other than DAAs Patients with sever heart failure or malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic hepatitis C virus patients will be on direct antiviral therapy attending to the outpatient clinics and inpatient of gastroenterology units of Internal medicine department .
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
glomerular filtration rate(eGFR) changes during HCV treatment | 3 month
  the frequency of renal impairment by evaluation of glomerular filtration rate(eGFR) changes during HCV treatment with direct antiviral drugs before and after the treatment using different equation for eGFR such as (MDRD, CKD_EPI,Cockroft)

SECONDARY OUTCOMES:
Effect of direct anti Viral drugs on kidney function | 3 month
  the frequency of renal impairment by direct antiviral drugs by measurement of serum BUN and creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Enas Alkareemy, MD, Study Director — Assuit university hospital

REFERENCES:
- [Background] Brown PR, Sadiq O, Weick A, Lenhart A, Elbatta M, Fernandez C, Kutait A, Pompa R, Jafri SM. Acute Kidney Injury in Patients Undergoing Chronic Hepatitis C Virus Treatment With Ledipasvir/Sofosbuvir. Hepatol Commun. 2018 Sep 24;2(10):1172-1178. doi: 10.1002/hep4.1243. eCollection 2018 Oct. PMID 30288472
- [Background] Soeiro CASP, Goncalves CAM, Marques MSC, Mendez MJV, Tavares APRA, Horta AMLMFCA, Sarmento-Castro RMDR. Glomerular filtration rate change during chronic hepatitis C treatment with Sofosbuvir/Ledipasvir in HCV/HIV Coinfected patients treated with Tenofovir and a boosted protease inhibitor: an observational prospective study. BMC Infect Dis. 2018 Aug 3;18(1):364. doi: 10.1186/s12879-018-3278-3. PMID 30075765
- [Background] Shah H, Bilodeau M, Burak KW, Cooper C, Klein M, Ramji A, Smyth D, Feld JJ; Canadian Association for the Study of the Liver. The management of chronic hepatitis C: 2018 guideline update from the Canadian Association for the Study of the Liver. CMAJ. 2018 Jun 4;190(22):E677-E687. doi: 10.1503/cmaj.170453. No abstract available. PMID 29866893